CLINICAL TRIAL: NCT06995651
Title: Pharmacokinetic and Pharmacodynamic Effects of Dorzagliatin in Pancreatic Insufficient-Cystic Fibrosis: A Randomized Double-blind, Cross-over Trial
Brief Title: Dorzagliatin in Pancreatic Insufficient Cystic Fibrosis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 858421
Record Dates: First submitted 2025-05-08; First posted 2025-05-29 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Insufficiency; Cystic Fibrosis-related Diabetes
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency | interventions — Dorzagliatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dorzagliatin (Experimental): Dorzagliatin 75 mg orally twice daily for 7 days
  Interventions: Drug: Dorzagliatin; Drug: Placebo
- Placebo (Placebo Comparator): matched-placebo orally twice daily for 7 days
  Interventions: Drug: Dorzagliatin; Drug: Placebo

INTERVENTIONS:
Drug: Dorzagliatin — Randomized, double-blind, cross-over study of Dorzagliatin 75 mg orally twice daily for 7 days compared to matched-placebo orally twice daily for 7 days.
Drug: Placebo — Randomized, double-blind, cross-over study of Dorzagliatin 75 mg orally twice daily for 7 days compared to matched-placebo orally twice daily for 7 days.

SUMMARY:
This study is designed to determine the pharmacokinetic and pharmacodynamic response of dorzagliatin 75 mg twice daily following 7-day administration in individuals with pancreatic insufficient cystic fibrosis and abnormal glucose tolerance when compared to randomized, double-blind 7-day administration of placebo in a cross-over fashion. We hypothesize that dorzagliatin administration will result in significant drug concentrations and improved glucose tolerance, early-phase insulin secretion, glucagon suppression, and hepatic glycogen storage assessed during a standardized mixed-meal tolerance test.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female, aged ≥18 years on date of consent.
4. Confirmed diagnosis of CF, defined by positive sweat test or CFTR mutation analysis according to CFF diagnostic criteria.
5. Pancreatic insufficiency defined by clinical requirement for pancreatic enzyme replacement.
6. Abnormal glucose tolerance defined by OGTT criteria for EGI, IGT, or CFRD, or diagnosed CFRD.
7. There will be no restriction on enrollment of individuals with CFRD but without fasting hyperglycemia (fasting hyperglycemia is defined as fasting glucose ≥126 mg/dL)

   a. Individuals with CFRD and fasting hyperglycemia (defined as above or by the use of basal insulin therapy) must also have a HbA1c ≤8% and a random (non-fasting) C- peptide ≥1.2 ng/mL [15].
8. For females of reproductive potential: use of highly effective contraception method for the during of study participation; oral contraceptives, intra-uterine devices, Norplant®, Depo- Provera®, and barrier devices with spermicide are acceptable contraceptive methods; condoms used alone are not acceptable.

Exclusion Criteria:

1. Established diagnosis of non-CF diabetes (e.g. type 1 diabetes).
2. Pregnancy or lactation; a negative urine pregnancy test will be required at enrollment.
3. Pulmonary exacerbation requiring IV antibiotics or systemic glucocorticoids within 4 weeks prior to randomization.
4. Treatment with either CYP3A4 inhibitors (e.g. ketoconazole, itraconazole, voriconazole, posaconazole, clarithromycin, indinavir, ritonavir, saquinavir, telithromycin, boceprevir, nelfinavir, telaprevir, conivaptan, nefazodone, etc.) or inducers (e.g. phenobarbital, other barbiturates, carbamazepine, phenytoin, rifampicin, dexamethasone, etc.).
5. Use of herbal remedies, including St. John's Wort within 14 days prior to dosing.
6. Change in CFTR modulator therapy in the previous 3 months.
7. History of clinically symptomatic pancreatitis within the last year.
8. Prior lung, liver or another solid organ transplant.
9. Abnormal kidney function: creatinine >2x upper limit of normal (ULN) or potassium >5.5mEq/L on non-hemolyzed specimen.
10. Abnormal liver function: persistent elevation of liver function tests >2.0 times ULN.
11. Uncontrolled hyperlipidemia: triglycerides >500 or cholesterol >250 mg/dl.
12. Hyperuricemia: serum uric acid >1.5 times ULN.
13. Anemia: hemoglobin <10 g/dL.
14. History of any illness or condition that, in the opinion of the investigator might confound the results of the study or pose an additional risk to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Drug concentrations (PK; Cmax) | 2 months
  Assessed by the peak glucose during a standardized mixed-meal tolerance test following 7-day administration of study drug
Glucose tolerance (PD) | 2 months

SECONDARY OUTCOMES:
Early-phase insulin secretion | 2 months
  Assessed by insulin secretory rate and
Glucagon suppression | 2 months
  Glucagon incremental area-under-the-curve (iAUC) analyses during the mixed-meal tolerance test following 7-day administration of study drug. iAUC analyses for GLP-1 and GIP will be assessed as potential effect modifiers.

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Rickels, MD, MS, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Hospital of University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pennsylvania Center for Human Phenomic Science (CHPS), Philadelphia, Pennsylvania